CLINICAL TRIAL: NCT04719572
Title: Intervention Study of Different Anti-osteoporpsis Intervention Strategies in Patients With Osteopenia and Osteoporosis
Brief Title: Intervention Study of Drugs in Patients Osteopenia and Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); Beijing Aerospace General Hospital (Other)
Responsible Party: Principal Investigator, Chunlin Li, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: antiosteoporosis301
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Osteoporosis; Osteopenia, Osteoporosis
Keywords: Anti-osteoporosis therapy; men; Postmenopausal women
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic treatment group (Other): elemental calcium 600mg/ day + vitamin D 1000IU/day
  Interventions: Other: Basic treatment+ anti-osteoporosis drug group; Other: Basic treatment + non-drug treatment group
- Basic treatment+ anti-osteoporosis drug group (Active Comparator): alendronate(70mg/week), zoledronate(5mg 1/ year), tripopeptide(20ug 1/day), denosumab(120mg/month), activated vitamin D(0.25ug 1/day), menatetrenone(15mg tid) according to the patient's condition
  Interventions: Other: Basic treatment group; Other: Basic treatment + non-drug treatment group
- Basic treatment + non-drug treatment group (Other): diet, exercise, rehabilitation therapy
  Interventions: Other: Basic treatment group; Other: Basic treatment+ anti-osteoporosis drug group

INTERVENTIONS:
Other: Basic treatment group — A total of 60 subjects were recruited in the group.
  Arms: Basic treatment + non-drug treatment group; Basic treatment+ anti-osteoporosis drug group
Other: Basic treatment+ anti-osteoporosis drug group — A total of 60 subjects were recruited in the group.
  Arms: Basic treatment + non-drug treatment group; Basic treatment group
Other: Basic treatment + non-drug treatment group — A total of 60 subjects were recruited in the group.
  Arms: Basic treatment group; Basic treatment+ anti-osteoporosis drug group

SUMMARY:
This is a 12 months, randomized, multicenter, open-label, parallel-group study in postmenopausal women and male aged 50 years or old with osteoporosis or osteopenia in China to evaluate the efficacy and safety of different anti-osteoporpsis intervention strategies.

DETAILED DESCRIPTION:
This is a 12 months,randomized, multicenter, open-label, pragmatic-group study in postmenopausal women and male aged 50 years or old with osteoporosis or osteopenia in China to evaluate the efficacy and safety of different anti-osteoporpsis intervention strategies, including

* Group1: Basic treatment group (elemental calcium 600mg/ day + vitamin D 1000IU/day)
* Group2: Basic treatment+ anti-osteoporosis drug group (alendronate, zoledronate, tripopeptide, denosumab, activated vitamin D, menatetrenone soft capsules according to the patient's condition)
* Group3: Basic treatment + non-drug treatment group(diet, exercise, rehabilitation therapy).

Eligibility for participation will be determined by medical history, physical examination, and laboratory results obtained during a screening visit. About 180 postmenopausal women and elderly male with osteoporosis or osteopenia will be included in this study.

All subjects will be given informed consent before starting any examination and test. The following data of all subject will be collected: liver and kidney function, HbA1c, fasting blood glucose, fasting lipid profile, serum calcium, serum phosphate, parathyroid hormone, 25-hydroxy vitamin D, bone turnover markers(BTMs) (inculding serum procollagen type I N-propeptide, serum C-terminal telopeptide of type I collagen,osteocalcin and alkaline phosphatase), thoracic and lumbar spine X-ray, bone mineral density(BMD) by dual energy X-ray.

Then they will be randomized into three groups at a 1:1 ratio. Every group will be given calcium carbonate and vitamin D. In the group 2, the medication will be decided by the doctor according to the patients' condition. Particularly, denosumab has not been approved for male adaptation, we will sign an additional informed consent.

All subjects will be followed by visiting clinic every three months and complete the examinations to assess the safety and efficacy. Safety indexes: liver and kidney function, urine routine test and 24-h urine calcium. Efficacy indexes: BMD change, BTMs changes and fracture reduction. All subjects will be followed 12 months and data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Postmenopausal women and male aged 50 years or old
* Osteoporosis by DXA or fragility fracture history
* Osteopenia with more than one osteoporotic risk factors

Exclusion Criteria:

* Secondary osteoporosis
* Renal insufficiency (Ccr< 35ml/min)
* New fractures < 3 months, prior bilateral hip fractures or surgical replacement.
* Other medication contraindications
* Malignant tumors
* Mobility-impaired individuals

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy on BTMs level | 3 months、6months、9months、12months
  The change of BTMs level after different interventions
The efficacy on BDM level | 12 months
  The change of BDM level after different interventions

SECONDARY OUTCOMES:
Fracture rate | 12 months
  Fracture rate during follow up
The type and rate of drug adverse reactions | 12 months
  The type and rate of drug adverse reactions during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Chunlin Li, M.D&Ph.D, Principal Investigator — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China